CLINICAL TRIAL: NCT05352685
Title: Effects of Propofol on Auditory Event-related Potentials and Brain Functional Connectivity in Patients With Supratentorial Glioma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Head of anesthesiology, Principal Investigator, Clinical Professor, Beijing Tiantan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: wxx19950421
Record Dates: First submitted 2022-04-18; First posted 2022-04-29 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Propofol; Glioma; Auditory Event-related Potential (AERP); Electroencephalogram (EEG); Brain Network Connectivity
MeSH Terms: conditions — Glioma | interventions — Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Active Comparator)
  Interventions: Drug: Propofol Injection
- supratentorial glioma patients (Experimental)
  Interventions: Drug: Propofol Injection

INTERVENTIONS:
Drug: Propofol Injection — 1% propofol is used for target-controlled infusion, and gradually increase the effect concentration at 0.2ug/ml. Make the subject's sedation depth reach light sedation and deep sedation respectively. EEG data were collected during wakefulness, light sedation, deep sedation, and recovery.

SUMMARY:
The growth of gliomas often infiltrates important brain tissues and impairs subcortical fiber transmission, resulting in changes in global brain network connectivity. Most of the current anesthesia depth monitoring methods are based on healthy brain function population，which is difficult to reflect the sedation depth of glioma patients accurately. Therefore, this study aims to explore the characteristics of brain network connectivity in glioma patients under different sedation depths by electroencephalogram (EEG) and auditory event-related potential (AERP) methods, which may provide a research basis for sedative titration and anesthesia depth identification in glioma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 60 years old;
2. American Society of Anesthesiologists (ASA) physical status rating I-II;
3. Supratentorial glioma (frontal, temporal, parietal, insular ；WHO grade I-III);
4. Native Chinese speaker;
5. Signed informed consent.

Exclusion Criteria:

1. Mallampati airway class≥III;
2. BMI>30kg/m2;
3. Combined OSAS or Stop-BANG score≥3;
4. Hearing impairment
5. Combined epilepsy symptoms
6. Recurrent or multiple intracranial tumors
7. Concomitant other psychiatric or neurological disorders
8. Pregnancy and lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The amplitude of auditory event-related potential | During the trial(up to 3 hours for each subject)
  The amplitude of MMN and P300
The latency of auditory event-related potential | During the trial(up to 3 hours for each subject)
  The latency of MMN and P300

SECONDARY OUTCOMES:
Brain network functional connectivity | During the trial(up to 3 hours for each subject)
  Using coherence ; phase slope index(PSI); phase locking value(PLV）;phase lag index(PLI）to evaluate the brain network functional connectivity of subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China